CLINICAL TRIAL: NCT05973890
Title: Community-based Communication Interventions for Increasing Repeat Donation Among First- Time Blood Donors in Ghana: A Pragmatic Type 1 Effectiveness- Implementation Hybrid Trial
Brief Title: Community-based Communication for Blood Donation in Ghana
Acronym: C-CAD
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); National Blood Service Ghana (Other); University of Ghana (Other); Syracuse University (Other); Liverpool School of Tropical Medicine (Other); University of Minnesota, Coordinating Centers for Biometric Research (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: B07; UH3HL151599-04 (NIH)
Record Dates: First submitted 2023-07-25; First posted 2023-08-03 (Actual); Last update posted 2025-07-14 (Actual); Status verified 2025-07

CONDITIONS: Increase Repeat Blood Donation Attempts Among First-time Donors

STUDY DESIGN:
Intervention Model Description: parallel 3 arm randomized controlled study with equal allocation
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- WhatsApp (Experimental): Participants assigned to the WhatsApp arm will receive messages, audios, images and videos in a moderated, closed WhatsApp group over a 14-month duration. The messages aim to motivate blood donation, encourage participants to discuss their blood donation experiences, and allow them to share their motivations for donating blood.
  Interventions: Behavioral: WhatsApp
- docudrama (Experimental): Participants randomized to this arm will meet three times (Month 2; Month 5 and Month 10), in a group setting, during the intervention. Each group will have a maximum of 20-40 participants. This is a stand-alone activity, which is not associated with a donation event. During each meeting, participants will be asked to watch, in the group setting, an episode of drama, lasting 15 minutes. The docudrama on blood donation will address participant's concerns regarding blood donation and address common donor fears.
  Interventions: Behavioral: docudrama
- control (No Intervention): standard of care for repeat blood donation

INTERVENTIONS:
Behavioral: WhatsApp — Participants assigned to the WhatsApp arm will receive messages, audios, images and videos in a moderated, closed WhatsApp group over a 14-month duration. The messages aim to motivate blood donation, encourage participants to discuss their blood donation experiences, and allow them to share their motivations for donating blood.
  Arms: WhatsApp
Behavioral: docudrama — Participants randomized to this arm will meet three times (Month 2; Month 5 and Month 10), in a group setting, during the intervention. Each group will have a maximum of 20-40 participants. This is a stand-alone activity, which is not associated with a donation event. During each meeting, participants will be asked to watch, in the group setting, an episode of drama, lasting 15 minutes. The docudrama on blood donation will address participant's concerns regarding blood donation and address common donor fears.
  Arms: docudrama

SUMMARY:
A randomized controlled trial to evaluate the effectiveness of the WhatsApp groups or docudrama compared to a control group (usual engagement with blood services) on repeat blood donation attempts among first-time blood donors in Ghana. Secondary outcomes will be blood donor retention, blood donation knowledge, attitudes, beliefs, motivations, intention to donate, and relatedness as potential mediators of blood donation behavior among first-time blood donors. The RCT will have three arms: 1. WhatsApp; 2. docudrama; 3. control. Each participant in the WhatsApp and docudrama arms will receive the intervention for 14 months. Participants in the control arm will receive standard national blood donation communications and be followed for 14 months. Actualized blood donation is possible every four months using NBSG guidelines; consequently, participants may make multiple blood donation attempts. Return blood donation attempts will be evaluated using the Southern Zonal Blood Center (SZBC) records (primary outcome) and participant self-report (secondary outcome) at 7 months and 14 months. Secondary measures will be evaluated at baseline, 7 and 14 months from enrollment. The duration of the RCT will be 26 months allowing for 12 months to achieve enrollment goals and 14 months of follow-up for the last individual enrolled.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years-old
* First-time whole blood donor with the SZBC of the NBSG
* Eligible to donate again at the time of eligibility confirmation
* Consent to participate
* Understands one of English, Twi, or Ga
* Have a smart phone
* Have, or be willing to sign up for an active WhatsApp account
* Be willing to watch a docudrama on blood donation in a group setting

Exclusion Criteria:

* History of more than one lifetime whole blood donation (with any blood center)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 882 (Actual)
Dates: Start 2024-01-15 (Actual); Primary Completion 2026-03-30 (Estimated); Study Completion 2026-03-30 (Estimated)

PRIMARY OUTCOMES:
Proportion with a repeat donation attempt | 14 months
  The primary outcome for the RCT will be the number of blood donation attempts

CONTACTS AND LOCATIONS:
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No
The BLOODSAFE project is committed to quickly sharing results and data. Papers will be submitted summarizing the primary results of the BLOODSAFE studies once the analysis is complete. These results will be published in major scientific journals and presented at scientific meetings.